CLINICAL TRIAL: NCT00411424
Title: Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Initial Efficacy of ASK8007 in Comparison With Placebo in Patients With Active Rheumatoid Arthritis - a Randomized, Double Blind, Placebo-controlled, Combined Single Dose Escalation and Multiple Dose Study
Brief Title: Safety, Tolerability and Efficacy Study of the New Medication ASK8007 to Treat Patients With Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8007-CL-0001; EudraCT number: 2006-000172-33
Record Dates: First submitted 2006-12-12; First posted 2006-12-14 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Randomized Control Trial; Treatment outcomes; Monoclonal antibody
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ASK8007 monoclonal antibody

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: ASK8007
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASK8007 — IV
  Arms: 1
Drug: Placebo — IV
  Arms: 2

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of the new medication ASK8007, and to study whether it has a beneficial effect on joint inflammation in patients with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* meet the American Rheumatism Association (ARA) 1987 revised criteria for the classification of RA (also referred to as the American College of Rheumatology [ACR] criteria);
* being treated with an adequate dose (to the discretion of the local physicians) of either MTX or leflunomide (LEF)or sulfasalazine (SS2) for at least 4 months prior to baseline of which the last 6 weeks before baseline were at a stable dose;
* have active poly-arthritis (i.e. active rheumatoid arthritis as defined in detail in the protocol)

Exclusion Criteria:

* have been treated with any registered or non-registered investigational drug in the context of a clinical intervention study during the last 3 months before baseline;
* have been treated with TNFα-blockers within a certain period of time (defined for each medication) before baseline;
* have been treated with any DMARD other than MTX, LEF or SS2 during the last month before baseline;
* documented evidence for the presence of clinically severe, unstable, or uncontrollable renal, hepatic, respiratory, hematological, genitourinary, cardiovascular, endocrine, neurological, psychiatric, or other medical illness which would, in the opinion of the investigator, put the patient at safety risk or mask measures of efficacy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability MD ASK8007 | up to 10 weeks after last dose

SECONDARY OUTCOMES:
DAS28+CD68 | Day 43 compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (10):
- Leuven, Belgium
- Budapest, Hungary
- Dublin, Ireland
- Netherlands (2):
  - Amsterdam
  - Groningen
- Spain (3):
  - A Coruña
  - Barcelona
  - Santiago
- United Kingdom (2):
  - London
  - Newcastle

REFERENCES:
- [Background] Boumans MJ, Houbiers JG, Verschueren P, Ishikura H, Westhovens R, Brouwer E, Rojkovich B, Kelly S, den Adel M, Isaacs J, Jacobs H, Gomez-Reino J, Holtkamp GM, Hastings A, Gerlag DM, Tak PP. Safety, tolerability, pharmacokinetics, pharmacodynamics and efficacy of the monoclonal antibody ASK8007 blocking osteopontin in patients with rheumatoid arthritis: a randomised, placebo controlled, proof-of-concept study. Ann Rheum Dis. 2012 Feb;71(2):180-5. doi: 10.1136/annrheumdis-2011-200298. Epub 2011 Sep 14. PMID 21917822